

# Clinical Development

# **EMA401**

### CEMA401A2202 / NCT03297294

A double-blind, placebo-controlled, randomized trial to determine the safety and efficacy of EMA401 100 mg b.i.d. in reducing 24-hour average pain intensity score in patients with painful diabetic neuropathy (EMPADINE)

# Statistical Analysis Plan (SAP)

Author: (CRO),

Document type: SAP Documentation

Document status: Amendment 1 Final

Release date: 18-Jun-2019

Number of pages: 36

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

# **Document History – Changes compared to previous final version of SAP**

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 16-<br>Feb-<br>2018 | Prior<br>to<br>FPFV | Creation of final version | N/A – First version | NA |
| 18-Jun-<br>2019 | Prior<br>to DB<br>lock | Creation of amendment 1 | Region names have changed. | 1.1, Study design,<br>, 2.5.2<br>Statistical, hypothesis,<br>model, and method of<br>analysis |
| | | | • modified FAS population has been added | 2.2. Analysis sets |
| | | | <ul> <li>vitals signs and Friderica's correction<br/>have been removed from demographic<br/>summary</li> </ul> | 2. 2.3 Patient disposition, demographics and other baseline characteristics |
| | | | analyses of prior and concomitant<br>medicationshave partly been revised and<br>described in more detail. Analyses<br>regarding prohibited medications have<br>been removed | 2.4 Treatments (study treatment, rescue medication, concomitant therapies) |
| | | | <ul> <li>supplementary analyses regarding the<br/>primary endpoint have been reduced. The<br/>second supplementary analysis has been<br/>kept</li> </ul> | 2.5 Analysis of primary objective |
| | | | covariate region has been removed from<br>the ANCOVA model | 2.7 Analysis of secondary efficacy |
| | | | <ul> <li>Tipping point analysis has been removed. A sensitivity analysis on the modified full analysis set has been added. </li> </ul> | objective(s) |
| | | | <ul> <li>Supplementary analyses of responders<br/>have been reduced. BPI-SF, PGIC, worst<br/>NRS, ISI will be summarized<br/>descriptively</li> </ul> | |
| | | | <ul> <li>Temporal items of NPSI will not be<br/>summarized descriptively. No summaries<br/>of the 5 dimensions of NPSI during the<br/>treatment withdrawal period will be<br/>provided</li> </ul> | 2.8.1 Adverse events (AEs) |

| Date | Time<br>point | Reason for update | | | on and title<br>cted (Current) |
|---|---|---|---|---|---|
| | | | <ul> <li>Analyses of AEs have been reduced. No<br/>subgroup analyses and analyses of drug-<br/>related AEs will be provided</li> </ul> | | |
| | | | • Dot plots and Kaplan Meier plots of AEs have been removed | 2.8.1.2 | Liver events |
| | | | | 2.8.3 | Laboratory data |
| | | | • Section has been removed. | 2.8.4 | Other safety data |
| | | | <ul> <li>Summary statistics of laboratory<br/>parameters, vital signs and ECG intervals<br/>will not be presented</li> </ul> | | |
| | | | Shift tables of laboratory data have been removed | | |
| | | | Bazett correction has been removed | | |
| | | | | 5.1.5 P<br>for PDS | rohibited medication S |
| | | | • For derivation of exclusion windows PD date can not be used | | |

| Та | | of conter | <b>nts</b><br>nts | 4 |
|---|---|---|---|---|
| | | | ations | |
| 1 | | | | |
| 1 | 1.1 | | lesign | |
| | 1.2 | , | objectives and endpoints | |
| 2 | | - | hods | |
| _ | 2.1 | | nalysis general information | |
| | | 2.1.1 | General definitions | |
| | 2.2 | | is sets | |
| | 2.3 | Patient | disposition, demographics and other baseline characteristics | |
| | | 2.3.1 | Patient disposition | |
| | 2.4 | | ents (study treatment, rescue medication, concomitant therapies, ance) | |
| | | 2.4.1 | Study treatment / compliance | 14 |
| | | 2.4.2 | Prior, concomitant and post therapies | |
| | 2.5 | Analysi | is of the primary objective | |
| | | 2.5.1 | Primary endpoint | 15 |
| | | 2.5.2 | Statistical hypothesis, model, and method of analysis | 16 |
| | | 2.5.3 | Handling of missing values/censoring/discontinuations | |
| | | 2.5.4 | Supportive analyses | 20 |
| | 2.6 | Analysi | is of the key secondary objective | 20 |
| | | 2.6.1 | Key secondary endpoint | 20 |
| | | 2.6.2 | Statistical hypothesis, model and method of analysis | 20 |
| | 2.7 | Analysi | is of secondary efficacy objective(s) | 21 |
| | | 2.7.1 | Responder Analysis | 21 |
| | | 2.7.2 | Other secondary efficacy objectives | 21 |
| | 2.8 | Safety a | analyses | 22 |
| | | 2.8.1 | Adverse events (AEs) | 22 |
| | | 2.8.2 | Deaths | 23 |
| | | 2.8.3 | Laboratory data | 24 |
| | | 2.8.4 | Other safety data | 25 |
| | 2.9 | Pharma | acokinetic endpoints | 26 |
| | 2.10 | PD and | PK/PD analyses | 26 |

| | 2.11 | Patient- | -reported outcomes | 26 |
|---|-------|------------|--------------------------------------------|----|
| | 2.12 | Biomar | rkers | 26 |
| | | | | 26 |
| | | | | 26 |
| | 2.14 | Interim | analysis - Safety | 27 |
| 3 | Samp | le size ca | alculation | 27 |
| 4 | Chan | ge to prot | tocol specified analyses | 28 |
| 5 | Appe | ndix | | 29 |
| | 5.1 | Imputa | tion rules | 29 |
| | | 5.1.1 | Study drug | 29 |
| | | 5.1.2 | Diagnosis of PDN | 29 |
| | | 5.1.3 | AE date imputation | 29 |
| | | 5.1.4 | Concomitant medication date imputation | 29 |
| | | 5.1.5 | Prohibited medication for PDN | 29 |
| | 5.2 | AEs co | oding/grading | 30 |
| | 5.3 | Labora | tory parameters derivations | 30 |
| | 5.4 | Derivat | tion of index values and scores | 30 |
| | | 5.4.1 | 11-point Numeric Rating Scale (NRS) | 30 |
| | | 5.4.2 | Verbal Rating Scale (VRS) pain intensity | 31 |
| | | 5.4.3 | Brief Pain Inventory- Short Form (BPI-SF) | 31 |
| | | 5.4.4 | Patient Global Impression of Change (PGIC) | 31 |
| | | 5.4.5 | Neuropathic Pain Symptom Inventory (NPSI) | 31 |
| | | 5.4.6 | Insomnia Severity Index (ISI) | 32 |
| | | | | 32 |
| | | | | 32 |
| | | | | 32 |
| | | | | 32 |
| | | | | 33 |
| | | 5.4.12 | Douleur Neuropathique 4 (DN4) | 34 |
| | 5.5 | Statistic | cal models | 35 |
| | | 5.5.1 | Primary analysis | 35 |
| | | 5.5.2 | Secondary analysis | 35 |
| | 5.6 | Rule of | f exclusion criteria of analysis sets | 35 |
| 6 | Refer | ences | | 36 |

Novartis For business use only Page 6 SAP CEMA401A2202

### List of abbreviations

ACR Albumin-Creatinine Ratio

AE Adverse Event
ALP Alkaline Phosphate

ALT Alanine Aminotransferase
ANCOVA Analysis of covariance

AST Aspartate Aminotransferase

ATC Anatomic Therapeutic Chemical classification

b.i.d. twice a day

BPI-SF Brief Pain Inventory-Short Form

CRO Contract Research Organization

CSR Clinical Study Report

DAR Dose Administration Record
DMC Data Monitoring Committee

DN4 Douleur Neuropathique en 4 Questions

ECG Electrocardiogram

eCRF Electronic Case Report Form

e-diary Electronic diary

EU European Union FAS Full Analysis Set

FDA Food and Drug Administration
GGT gamma-glutamyltransferase

HIV Human Immunodeficiency Virus

INR International Normalized Ratio
IRT Interactive Response Technology

ISI Insomnia Severity Index

J2R Jump to reference
LFT Liver function test
LoE Lack of efficacy
MAR Missing at random

mFAS Modified Full Analysis Set

MedDRA Medical dictionary for regulatory activities
NPSI Neuropathic Pain Symptom Inventory

NRS Numeric Rating Scale

NSAID Nonsteroidal Anti-inflammatory Drugs

PCR Protein-Creatinine Ratio
PDN Painful Diabetic Neuropathy

| Novartis | For business use only | Page 7 |
|----------|-----------------------|--------------|
| SAP | | CEMA401A2202 |

| PHN | Post-Herpetic Neuralgia |
|------|----------------------------------------|
| PK | Pharmacokinetics |
| PGIC | |
| | Patient Global Impression of Change |
| PRO | Patient Reported Outcome |
| QTc | Corrected QT interval |
| QTcB | Bazett QT correction formula |
| QTcF | Fridericia QT correction formula |
| SAE | Serious Adverse Event |
| RDO | Retrieved drop-out |
| SAF | Safety population |
| SSRI | Selective Serotonin Reuptake Inhibitor |
| TBL | Total bilirubin |
| TD | Study Treatment Discontinuation |
| TEAE | Treatment-Emergent Adverse Events |
| ULN | Upper limit of Normal |
| USM | Urgent Safety Measures |
| VRS | Verbal Rating Scale |
| WHO | World Health Organization |

#### **Amendment 1**

This amendment of the statistical analysis plan (SAP) is largely based on changes induced due to the early termination of the CEMA401A2202 study. 137 patients out of 400 planned patients have been randomized. As the number of patients included in the study isconsiderably reduced, an abbreviated Clinical Study Report (CSR) that still meets all requirements for reporting and disclosure of the demographics, primary endpoint, secondary endpoints and safety results to public registries will be created.

The primary analysis on the change from baseline to Week 12 in the weekly mean of the 24-hour average pain score will be performed as originally planned. Besides the primary estimand, which is of main clinical interest, the supplementary estimand, which provides insight into the magnitude of improvement in efficacy that might be achieved if all patients were able to take EMA401 as prescribed for 12 weeks, will be analysed. The other planned supplementary estimands will be dropped, as they are of minor interest in the situation with many study treatment discontinuations due to trial termination in the scope of the Urgent Safety Measures (USM).

To support the primary analysis and to get an idea about the effect that might be achieved if the trial had not been terminated and if all patients had the chance to complete the Week 12 assessment, a sensitivity analysis on a modified population will be performed. The modified full analysis set will include all patients who had a chance to complete the study before the termination date, i.e who had been randomized at least 12 weeks before study termination date.

Similar considerations were made for the key-secondary endpoint.

Due to the considerably reduced number of patients who completed the study, only descriptive subgroup analyses will be provided. Moreover, the secondary endpoints will also be summarized descriptive only.

### 1 Introduction

This statistical analysis plan (SAP) describes all planned analyses for the Clinical Study Report (CSR) of study CEMA401A2202, a Phase 2, double-blind, placebo-controlled, randomized trial to determine the safety and efficacy of EMA401 in reducing 24-hour average pain intensity score in patients with painful diabetic neuropathy.

The content of this SAP is based on the final version of protocol CEMA401A2202 (release date 15-Sep-2017). All decisions regarding final analysis, as defined in the SAP document, have been made prior to database lock and unblinding of the study data.

# 1.1 Study design

The study is interventional, randomized, parallel, placebo-controlled, double-blind treatment.

The study will consist of a Screening epoch (up to 4 weeks), a double-blind Treatment epoch (12 weeks), and a double-blind Treatment withdrawal epoch (1 week).

• Patients will be randomized in a 1:1 ratio to treatment with placebo or EMA401 100 mg b.i.d.

Overall approximately 400 patients will be enrolled in the study (i.e. approximately 200 patients will be enrolled in each treatment arm).

At Week 12 (Visit 199), all patients who completed the 12-week double-blind Treatment epoch will enter the 1-week double-blind Treatment withdrawal epoch. The IRT system will indicate the unique medication number for the package of study drug to be dispensed to the patient during the double-blind Treatment withdrawal epoch. This medication number will correspond to the blinded withdrawal regimen assigned at Baseline.

Randomization will be stratified by region (America, Europe and Australia) and use of concomitant pain medication for PDN (yes/no) in order to achieve balance of treatment allocation within the stratification factors.

Primary objective of this study is to compare the efficacy of EMA401 vs. placebo in 24-hour average pain intensity score at Week 12, using an 11 point Numeric Rating Scale (NRS) by testing the superiority of EMA401 100 mg b.i.d. vs. placebo.

## 1.2 Study objectives and endpoints

Table 1-1 Objectives and related endpoints

| Objective(s) | Endpoint(s) |
|---|---|
| Primary Objective(s) To compare the efficacy of EMA401 vs. placebo in 24-hour average pain intensity score at Week 12, using an 11 point Numeric Rating Scale (NRS) by testing the superiority of EMA401 100 mg b.i.d. vs. placebo | Change in weekly mean 24-hour average pain score (using the 11 point NRS) from Baseline to Week 12 |
| Key Secondary Objective(s) | Endpoint(s) for key secondary objective(s) |

#### Objective(s)

#### To compare the efficacy of EMA401 vs. placebo in Neuropathic Pain Symptom Inventory (NPSI) total score by testing the superiority of EMA401 100 mg b.i.d. vs. placebo

#### Endpoint(s)

 Change in Neuropathic Pain Symptom Inventory (NPSI) total score from Baseline to Week 12

#### Secondary Objective(s)

#### To evaluate the efficacy of EMA401 compared to placebo, as measured by the Brief Pain Inventory-Short Form (BPI-SF) interference total score at Week 12

- To evaluate the efficacy of EMA401 compared to placebo, as measured by the weekly mean of the 24-hour worst pain intensity score, using an 11-point Numeric Rating Scale (NRS) at Week 12
- To evaluate the efficacy of EMA401 compared to placebo, on the Patient Global Impression of Change (PGIC) at Week 12
- To evaluate the proportion of EMA401 patients achieving a ≥ 30% and a ≥ 50% reduction in weekly mean 24-hour average pain intensity score using the NRS compared to placebo (i.e., responder rates) at Week 12
- To evaluate the effect of EMA401 compared to placebo on the Insomnia Severity Index (ISI) at Week 12
- To evaluate the safety and tolerability of EMA401 compared to placebo in PDN patients, as measured by treatment emergent adverse events (TEAEs), adverse events (AEs) leading to study drug discontinuation and serious adverse events (SAEs) throughout the study
- To evaluate the pharmacokinetics (PK) of EMA401 and exposure-response (decrease in pain intensity) relationship for EMA401 throughout the study
- To evaluate the proportion of patients who need rescue medication separately for the double-blind Treatment epoch and Treatment withdrawal epoch an the time first intake of rescue medication during the double-blind Treatment epoch.

#### Endpoint(s) for secondary objective(s)

- Change in BPI-SF interference total score from Baseline to Week 12
- Change in weekly mean of the 24-hour worst pain score, using an 11-point NRS, from Baseline to Week 12
- PGIC at end of study
- Proportion of patients meeting responder criteria from Baseline to Week 12
- Change in ISI from Baseline to Week 12
- Number and severity of treatment emergent adverse events and the frequency of adverse events leading to discontinuation. Number of serious adverse events.
- Plasma pharmacokinetics of EMA401 will be characterized by population nonlinear mixed effects modeling techniques
- Proportion of patients who need rescue medication separately for the doubleblind Treatment epoch and Treatment withdrawal epoch, the time to first intake of rescue medication during the doubleblind Treatment epoch



## 2 Statistical methods

# 2.1 Data analysis general information

The statistical analysis of the study will be performed by Contract Research Organization (CRO).

SAS version 9.4 will be used to perform all data analyses and to generate tables, figures and listings.

Qualitative data (e.g., gender, race, etc.) will be summarized by means of frequency tables; a missing category will be included as applicable. Percentages will be calculated using the number of patients in the relevant population or subgroup as the denominator.

Quantitative data (e.g., age, body weight, etc.) will be summarized by appropriate descriptive statistics, i.e., n, mean, standard deviation (SD), first quartile (Q1), median, third quartile (Q3), minimum, and maximum.

No interim analysis will be performed for the efficacy evaluation. An external Data Monitoring Committee (DMC) will be established with the primary goal to perform an ongoing review of safety data.

#### 2.1.1 General definitions

#### Investigational drug and study treatment

The investigational drug, EMA401, will be provided as capsules. The following oral dosage strengths will be used: 50 mg.

EMA401 and placebo will be identical in appearance.

For all treatment groups, each dose will be self-administered orally as two capsules with a full glass of non-carbonated water twice daily, consisting of a morning dose and an evening dose.

The following abbreviated treatment groups, independently of cohort number, will be used as the headers in the tables for the double-blind Treatment epoch:

- Placebo b.i.d.
- EMA401 100 mg b.i.d.

The following abbreviated treatment groups will be used as the headers in the tables for the double-blind Treatment withdrawal epoch:

- Placebo b.i.d. -> Placebo b.i.d.
- EMA401 100 mg b.i.d. -> EMA401 100 mg b.i.d.
- EMA401 100 mg b.i.d. -> Placebo b.i.d.

## Date of first and last administration of study drug

The date/time of first administration of study drug is defined as the first date/time of administration as per Dosage Administration Record eCRF. The date/time of last administration of study drug is defined as the last date/time when a dose is administered as per Dosage Administration Record eCRF. This value has to be compared to the "End of study treatment" as recorded on the corresponding eCRF. In case of different dates, the latest will be used as treatment end.

For subjects with missing first dose date, the randomization date will be considered as reference start date.

## Study day

The study day, describes the day of the event or assessment date, relative to the reference start date which is the date of first administration of study drug.

The study day is defined as:

- The date of the event (visit date, onset date of an event, assessment date etc.) reference start date + 1 if event is on or after the reference start date.
- The date of the event (visit date, onset date of an event, assessment date etc.) reference start date if event precedes the reference start date.

#### Baseline

For safety and efficacy evaluations, the last available assessment (either scheduled or unscheduled) before the first administration of study drug and after the screening visit is defined as "baseline" assessment. If patients have no value prior to first administration of study drug the baseline result will be missing.

#### Post-baseline

For safety and efficacy evaluations all assessments after the first administration of study drug are defined as "post-baseline" assessment.

## Change and percent change from baseline for continuous parameter.

Change from baseline and percent change from baseline will only be summarized for subjects with both baseline and post-baseline values and will be calculated as:

change from baseline = post-baseline value – baseline value

percent change from baseline = 100 \* change from baseline / baseline value.

For summary statistics the raw values (and not imputed values) will be used.

#### Study periods and date of last contact

The overall observation period will be divided into three mutually exclusive segments:

- A screening phase of up to 4 weeks
- A double-blind treatment phase starting with first dose of study drug at Visit 101 and covering 12 weeks of treatment.
- A double-blind treatment withdrawal phase for one week starting after 12 weeks of treatment with Visit 201.

Inferential analysis will be performed on either only treatment phase or on both treatment and treatment withdrawal phase separately. It is never the case that both phases will be pooled together.

#### Visit windows

| Visit win | dows will b | oe applie | ed for all | meası | ureme | ents except | NRS sc | ores. The d | efinition of |
|---|---|---|---|---|---|---|---|---|---|
| seamless | windows | can b | e found | in | the | following | | location | |
| | | | | The r | nost | recent versi | ion of tl | his documer | nt available |
| before the | database 1 | ock will | be used t | o det | ermin | e the visit | window | s for baseling | ne and post |
| baseline v | isits and tre | atment d | liscontinua | tion v | isit n | napping. | | | |

# 2.2 Analysis sets

The following analysis populations will be used for analysis.

- The Enrolled population will include all patients who were enrolled into the study.
- The Full Analysis Set (FAS) comprises all patients to whom the study treatment has been assigned. Following the intention-to-treat principle, patients will be analyzed according to the treatment assigned to at randomization. Mis-randomized patients will be excluded from the FAS.
- The modified Full Analysis Set (mFAS) will include all patients who could have completed Week 12 by the study termination date. That means, all patients which were randomized at least 12 weeks prior to 25-Feb-2019 will be included.
- The Safety population (SAF) will include all patients who took at least one dose of study medication. Patients will be analyzed according to treatment received.

The primary efficacy analysis will be performed on the FAS.



# 2.3 Patient disposition, demographics and other baseline characteristics

Patient demographic and baseline characteristic data to be collected on all patients include: year of birth, age, sex, race, ethnicity, relevant medical history/current medical condition present before signing informed consent, height, weight, body mass index (BMI), prior concurrent medications, NRS at screening,

In addition, the following categorizations of continuous variables will be done:

- Age into 18-64 years, 65-84 years, >= 85 years;
- Duration of PDN into < 1 year, > 1 5 years, > 5 10 years, > 10 15 years, > 15 20 years, and > 20 years;

Duration of PDN is calculated from the start date of PDN as reported on the eCRF until the date of Visit 1.

Demographic and background information will be summarized the FAS population using frequency distributions (for categorical variables) and descriptive statistics of mean, standard deviation, minimum, median and maximum (for continuous variables). Relevant medical history/current medical conditions will be summarized by system organ class and preferred term of the MedDRA dictionary.

#### 2.3.1 Patient disposition

For each study phase (i.e., Screening, Treatment epoch and Treatment withdrawal epoch), the overall number of patients who entered, completed, and discontinued that phase will be summarized including the reasons for discontinuation. The summary of the screening phase will be done for the Enrolled set, for the Treatment and Treatment withdrawal epoch. The analyses will be based on the FAS population.

Patients who prematurely discontinue the study medication will be listed along with the reasons for discontinuation.

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

## 2.4.1 Study treatment / compliance

Duration (days) of exposure to double-blind study medication will be summarized by treatment group and treatment phase (Treatment epoch and Treatment withdrawal epoch seperately). In addition, the number of subjects with exposure of at least certain time thresholds (any exposure, >= 1 week, >= 2 weeks, >= 4 weeks, >= 6 weeks, >= 8 weeks, >= 10 weeks, >= 12 weeks) will be displayed.

Compliance will be recorded as source documentation only and not analysed.

The analyses will be based on the SAF population.

## 2.4.2 Prior, concomitant and post therapies

The number and percentage of patients who used concomitant medications (coded by World Health Organization [WHO] Anatomic Therapeutic Chemical classification [ATC]) will be presented by treatment group and treatment phase (Treatment epoch and Treatment withdrawal epoch separately).

Separate tabulations will be provided for medications taken prior to start of study medication and while a patient is on study drug (i.e. concomitant, between the first day on study drug and the day of last visit). In addition, the PDN medications recorded on the Screening PDN Medication Log will be summarized using a frequency table for each medication. The primary reason for treatment failure will also be tabulated.

Prior medications are defined as drugs taken and stopped prior to first dose of study treatment. For the Treatment epoch concomitant medications are defined as any medication given at least once between the day of first dose of study treatment and the end of the treatment epoch, including those which were started pre-baseline and continued into the treatment period. For the Treatment withdrawal epoch concomitant medications are any medications given at least once between the day of first dose of study medication in the treatment withdrawal epoch, and the end of the epoch, including those which were started pre-baseline or in the treatment period epoch, and continued into the treatment withdrawal epoch.

Non-drug therapies will be listed.

#### 2.4.2.1 Rescue medication

The number and percentage of patients who received rescue medication (Acetaminophen/Paracetamol as reported on the diary page) will also be summarized by treatment and by visit during the double-blind treatment and treatment withdrawal period separately. Visit mapping will be done according to the visit window strategy document (see Section 2.1.1). The dose received will be listed.

Analysis of time to first use of rescue medication will be performed using Kaplan-Meier curves.

Number of patients with at least one intake will also be summarized.

# 2.5 Analysis of the primary objective

#### 2.5.1 Primary endpoint

The primary efficacy variable will be the change from baseline to Week 12 in the weekly mean of the 24-hour average pain score, using an 11-point Numeric Rating Scale (NRS).

The NRS is captured in the e-diary daily by the patient as the intensity of pain in the past 24 hours. To calculate the weekly mean pain intensity score for a given week, the daily pain

intensity scores collected by the patient in the e-diary during the 7 days of that week will be averaged.

The primary population will be the FAS.

## 2.5.2 Statistical hypothesis, model, and method of analysis

The aim is to estimate the treatment effect of the investigational drug (EMA401) compared to placebo, for the target population on the primary pain parameter. The definition and the justification of the corresponding primary estimand, as well as the definition of the supplementary and secondary estimands for NRS are detailed in the Estimand Charter. The most recent version of the Estimand charter stored at

available before the database lock will be used as reference.

The primary estimation method is based on an Analysis of Covariance (ANCOVA) model including treatment, sex, use of concomitant pain medication for PDN (yes/no) as factors and age and baseline (mean pain intensity) score as covariate. The analysis will account for different intercurrent events (i.e. events that occur post-randomization) as follows:

- Changes in doses of concomitant medication for PDN: Efficacy observations collected during the period of changes in doses of concomitant medication for PDN (compared to baseline) and the 3-days thereafter will be excluded, since they are considered affected by the concomitant medication dose change. The resulting missing data after this step will be imputed via multiple imputation method using the Missing at random (MAR) assumption.
- **Intake of rescue medication:** Efficacy data collected during intake of rescue medication will be used for analysis.
- Intake of prohibited medications with potential confounding effect prior to study treatment discontinuation: The prohibited medications with a potential confounding effect are defined as those listed in Table 2-1 requiring study treatment discontinuation. A list of prohibited medications is available at the following

. Efficacy observations collected during the intake period of such prohibited medications and the 7-days thereafter will be excluded, since they are considered affected by the prohibited medication intake. The resulting missing data after this step will be imputed via multiple imputation method using the MAR assumption.

Table 2-1 Prohibited medication

| Medication | Prohibition period | Action taken for study treatment |
|---|---|---|
| Prohibited prior to Screening and throughout study | | |
| Any skeletal muscle relaxant (e.g. baclofen, orphenadrine, methocarbamol) | 2 weeks prior to Screening and after Screening | None |
| Mexiletine | 2 weeks prior to Screening | None |

| Medication | Prohibition period | Action taken for study treatment |
|---|---|---|
| | and after Screening | |
| Dextromethorphan | 2 weeks prior to Screening and after Screening | None |
| Memantine | 2 weeks prior to Screening and after Screening | None |
| Alpha-lipoic acid | 2 weeks prior to Screening and after Screening | None |
| Other anti-epileptic drugs (e.g. valproic acid, carbamazepine, phenytoin) | 2 weeks prior to Screening and after Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Antiviral medications (e.g. valacyclovir, acyclovir, amantadine, anti-HIV) | 2 weeks prior to Screening and after Screening | None |
| High dose capsaicin patch (8%) | 6 months prior to Screening and after Screening | Discontinue study treatment |
| Prohibited after Screening and through | nout study | |
| Oral or injectable steroids | After Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Monoamine oxidase inhibitors or any other antidepressants (except stable dosage of SSRI) | After Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Antipsychotic or neuroleptic medications | After Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Cannabinoids (e.g. marijuana) | After Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Prescribed opioids, including codeine | After Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Prescription systemic pain medication, or <i>topical</i> treatment for PDN, including lidocaine plaster | After Screening | Discontinue study treatment upon 2 <sup>nd</sup> episode of medication use |
| Nonsteroidal Anti-inflammatory Drugs (NSAIDs) or any other over-the-counter pain medications | After Screening | None |
| Any non-drug therapies that could modulate the perception of pain either directly or indirectly (i.e. transcutaneous electrical nerve simulation (TENS) or surgery) | After Screening | Discontinue study treatment |

| Medication | Prohibition period | Action taken for study treatment |
|---|---|---|
| Other medications that may have potential drug-drug interactions (e.g. felodipine, eplerenone, nisoldipine, ticagrelor, tacrolimus, avasimibe, rifampin, cyclosporine, gemfibrozil, clarithromycin, St. John's Wort; oral, injected or implanted hormonal methods for contraception) | After Screening | None |

Retrieved drop-out (RDO) patients are defined as patients who discontinue study treatment and decide to remain in the study by following an abbreviated schedule of assessments. These patients must continue to adhere to protocol requirements (see respective protocol Table 6-2). The design feature of retrieved drop-outs, considered in order to minimize the occurrence of missing data on primary pain parameter, is exploited for the statistical analysis as follows:

- Permanent discontinuation of study treatment due to AE, lack of efficacy (LoE) and use of prohibited medication: If retrieved drop-out data are available, these will be used for analysis. If no data was retrieved after study treatment discontinuation, missing data will be multiply imputed based on placebo arm data, i.e. "jump to reference" (J2R) assumption for the EMA401 arm, missing at random assumption for placebo arm (Carpenter, Roger, and Kenward 2013). Of note, alternatively one could build the imputation model based on the RDO data, however, we expect sparse RDO data which will likely hinder us to build an imputation model. More details on the imputation model are specified in Section 5.
- Permanent discontinuation of study treatment due to other reasons than AE, LoE and use of prohibited medication (including discontinuation due to USM): If efficacy data collected after study treatment discontinuation are available (retrieved drop-out), then the retrieved drop-out data will be excluded and missing data after study treatment discontinuation will be imputed via multiple imputation method using the MAR assumption.

The multiple imputations will be carried out on the weekly mean pain score. Details on multiple imputation can be found in Section 5 of this document.

The primary objective will be achieved if the EMA401 100 mg b.i.d. dose is statistically significant versus placebo in terms of the primary efficacy variable after multiplicity adjustment. To preserve the family-wise error rate at 2.5% level when comparing the EMA401 100 mg b.i.d. dose versus placebo on the primary and key secondary endpoints (see Section 2.6), statistical testing will be carried out using the following sequentially rejective, weighted Bonferroni-type test using the graphical approach (Bretz et al 2009) mentioned in Figure 2-1.

Figure 2-1 Sequentially rejective, weighted Bonferroni type test using the graphical approach



In the graphical testing procedure given in Figure 2-1, H1 and H2 denote the two null hypotheses of no treatment difference of EMA401 100 mg b.i.d. vs. placebo for the primary efficacy variable NRS and key secondary efficacy variable NPSI total score. The corresponding alternative hypotheses will be EMA401 100 mg b.i.d. is superior to placebo for the NRS and NPSI respectively. In the Figure 2-1 the number in the circle represents the proportion of alpha level to be assigned at the initial stage among the two null hypotheses. The direction and the number in the arrow represent the proportion of the alpha to be propagated to the next hypothesis. Initially, H1 will be tested at the full alpha level (1 sided) 0.025. If H1 is rejected then H2 will be tested also at the full alpha level (1 sided) 0.025.

To facilitate the interpretation of the estimated treatment difference a standardized effect size will be provided and will be calculated based on the results of the ANCOVA analysis.

The same ANCOVA model will be applied at the visits prior to Week 12. Multiplicity adjustment at visits prior to Week 12 will not carried out.

Summary statistics for absolute values and change from baseline by treatment and visit will be provided for the original measurements (i.e. for the raw data prior to multiple imputation) of the primary efficacy variable. If a measurement is collected under the period of use of prohibited medications or the 7 days thereafter, it will be excluded from the summaries.

## 2.5.3 Handling of missing values/censoring/discontinuations

#### Handling of missing daily pain score values within a week (within-week imputation)

The 24-hour average pain score is measured daily for seven consecutive days prior to randomization and then every day through the end of the study. At each week, the weekly mean of the seven 24-hour average pain assessments will be calculated.

The weekly mean will be calculated based on the available assessments. If only one measurement is available, the mean will be based on that value. Assessments made under treatment will not be mixed up with RDO data. If there is at least one value among the seven values in one week which is on-treatment, the mean will be calculated based on that.

#### Handling of missing weekly mean pain score values (weekly mean imputation)

The multiple imputation for the primary variable will be carried out on the weekly mean pain score.

The imputation procedure related to primary analysis is described in Section 2.5.2 while the imputation procedure for the supplementary analyses is included in Section 2.5.4. The details of these imputation rules are specified in the Estimand Charter and in Section 5.

For all analyses, imputation of intermittent missing observations before treatment discontinuation will be carried out following a MAR mechanism for all treatment arms.

# 2.5.4 Supportive analyses

## 2.5.4.1 Supplementary analysis

The following supplementary analysis to the primary analysis for NRS will be performed on the FAS population.

to quantify the treatment effect of the investigational drug compared to placebo, that would have been observed had all patients remained on their assigned treatment for 12 weeks. The handling of post randomization events will be same as for the primary analysis, except that missing data after discontinuation for any reason will be imputed using the MAR assumption.

The supplementary estimand corresponding to this supplementary analysis is described in detail in the Estimand Charter.

#### 2.5.4.2 Sensitivity analysis

A sensitivity analysis will be performed on the mFAS population using the same ANCOVA model as for the primary analysis.

## 2.6 Analysis of the key secondary objective

# 2.6.1 Key secondary endpoint

The key secondary efficacy variable will be the change from baseline to Week 12 in the Neurophathic Pain Symptom Inventory (NPSI) total score which is calculated as the sum of 10 descriptors outcome measure out of the 12 items measured in the NPSI.

The key secondary endpoint will be evaluated for the FAS.

## 2.6.2 Statistical hypothesis, model and method of analysis

To compare the efficacy of EMA401 over placebo in the NPSI total score the null hypothesis of superiority of EMA401 over placebo will be tested. The definitions of the estimands for the key secondary variable NPSI will also be detailed in an Estimand Charter.

The estimation of the treatment difference and missing data handling will be performed using the method of analyses mentioned for the primary analysis for NRS. Post randomization events will be handled in the same way as in the primary analysis for NRS.

The key secondaray objective will be achieved if the EMA401 100 mg b.i.d. dose is statistically significant versus placebo in terms of NPSI total score after multiplicity adjustment. To preserve the family-wise error rate at the 2.5% level when comparing the EMA401 100 mg b.i.d. dose versus placebo on the two endpoints NRS and NPSI, statistical testing will be carried out using the graphical testing procedure as explained in Section 2.5.2.

The same ANCOVA model will be applied at the visits prior to Week 12. Multiplicity adjustment at visits prior to Week 12 will not carried out.

The same supplementary analysis as for the primary endpoint will be performed.

Summary statistics by treatment and visit will be provided for the key secondary endpoint.

# 2.7 Analysis of secondary efficacy objective(s)

The following secondary efficacy variables will be evaluated for the FAS:

## 2.7.1 Responder Analysis

Responder analyses (based on at least a 30%, 50% improvement from baseline on NRS) will be performed in order to facilitate the interpretation of the results of the primary and supplementary analysis from a clinical relevance perspective. These analyses will be performed on the FAS population. One secondary estimand is considered, together with one supplementary estimand.

The secondary estimand and the supplementary estimand to the secondary estimand differ from the primary and supplementary estimand in two ways:

- First, the variable of interest is the responder status in NRS score, with response status corresponding to at least a 30% (50%) improvement in pain from baseline.
- Second, the measure of intervention effect is the odds ratio of the proportions of responders between investigational drug and placebo.

The other features characterizing these responder analyses are exactly the same as for the primary and the t supplementary analysis, respectively.

From an analysis point of view, the responder status for each patient will be calculated on the continuous weekly score measurements after missing data are multiply imputed based on the approach specified corresponding to the primary analysis and the supplementary analyses. If the patient is a completer but week 12 measurement is affected by the changes in doses of concomitant medication for PDN or the use of prohibited medication then the responder criteria will be defined based on the multiply imputed values by MAR. The resulting responder variable will be analyzed using a logistic regression model including all randomized patients and adjusting for the same covariates as the ANCOVA model for the primary analysis.

From an analysis point of view, the resulting responder variables will be analyzed using a logistic regression model including all randomized patients (FAS population) and adjusting for the same covariates as the ANCOVA model for the primary analysis. Odds ratios will be estimated along with their 95% CIs.

The responder analyses will be performed for each visit, with the obvious modification in the definition for the week of interest.

# 2.7.2 Other secondary efficacy objectives

- 1. BPI-SF interference total score will be summarized descriptively by treatment and visit...
- 2. Weekly mean of the 24-hour **worst** NRS pain score, using an 11-point Numeric Rating Scale (NRS). This variable will be summarized descriptively by treatment and visit.

- 3. Number of patients in each level of PGIC at end of study treatment will be presented by treatment. PGIC classification will also be combined into two categories: Either a "very much improved" or a "much improved" reported, and the five remaining categories.
- 4. Insomnia Severity Index (ISI) will be summarized descriptively by treatment and visit.
- 5. The proportion of patients who need rescue medication (at each visit and at least once during the study) will be evaluated separately for the double-blind Treatment epoch and Treatment withdrawal epoch.
- 6. The Kaplan-Meier estimates of the proportion of patients with rescue medication intake during the double-blind Treatment epoch, along with the associated 95% confidence intervals using the Greenwood's formula will be provided.

# 2.8 Safety analyses

Safety analyses will be conducted using the safety (SAF) population. Patients will be analysed by the actual treatment they received. All the safety analyses including AEs, vital signs, laboratory parameters, ECGs will be reported for double-blind treatment period as well as for the treatment withdrawal period separately.

## 2.8.1 Adverse events (AEs)

Treatment-emergent adverse events (TEAEs) are defined as any adverse events that develops after initiation of study treatment until the end of study visit or any event already present that worsens following exposure to the study treatment.

If an adverse event starts at the date of week 12 visit it should be allocated to the treatment epoch and not to the treatment withdrawal epoch. Adverse events reported 21 days after end of study date in the scope of USM will not be included in the summary tables, but will be listed.

TEAEs will be summarized (number of cases as a percentage of number at risk) by treatment group separately for Treatment epoch and Treatment withdrawal epoch. Number and percentage of patients with TEAE will be summarized by primary system organ class and preferred term for each treatment group during the double-blind Treatment epoch and during the double-blind Treatment withdrawal epoch. Severity will be classified as "mild", "moderate" and "severe". Serious TEAEs, TEAEs by maximum severity and TEAEs leading to premature discontinuation from study drug will be presented in a similar format as adverse events. Additionally, a listing of patients with TEAE will be presented. Drug abuse-related adverse events (identified using a pre-specified search criterion) will be summarized during the double-blind Treatment epoch. To assess the potential for withdrawal effect, drug abuse-related adverse events will be summarized for the double-blind Treatment withdrawal epoch.

The following additional analysis will be performed.

• Analysis of treatment-emergent adverse events with onset date before 25-Feb-2019

For rash adverse events, following details will be listed:

• Laterality and location of rash

- Did the subject start any new topical non-pharmaceutical products within the last 14 days prior to the start of rash?
- Topical Non-pharmaceutical Products related to the event of rash including soap, detergent, perfume, cologne and lotion.
- Were there any additional contributing factors that may have led to the rash?
- Did the dermatologist agree with the event?
- Additional investigation performed to diagnose that event: yes, no

For the legal requirements of ClinicalTrials.gov and EudraCT, two required tables on <ontreatment/treatment emergent> adverse events which are not serious adverse events with an incidence greater than X% and on <on-treatment/treatment emergent> serious adverse events and SAE suspected to be related to study treatment will be provided by system organ class and preferred term on the safety set population.

If for a same patient, several consecutive AEs (irrespective of study treatment causality, seriousness and severity) occurred with the same SOC and PT:

- a single occurrence will be counted if there is  $\leq 1$  day gap between the end date of the preceding AE and the start date of the consecutive AE
- more than one occurrence will be counted otherwise.

For occurrence, the presence of at least one SAE / SAE suspected to be related to study treatment / non SAE has to be checked in a block e.g., among AE's in a  $\leq$  1 day gap block, if at least one SAE is occurring, then one occurrence is calculated for that SAE.

The number of deaths resulting from SAEs suspected to be related to study treatment and SAEs irrespective of study treatment relationship will be provided by SOC and PT.

#### 2.8.1.1 Adverse events of special interest / grouping of AEs

Allergic dermatitis, elevation in hepatic enzymes and neutropenia are the potential risks related to EMA401. Dizziness, headache, nausea, pre syncope and upper respiratory tract infections are the expected events related to EMA401. In addition suicidality and drug abuse related events will be adverse events of special interest. The search criterion for each of these risks and events will be defined based on MedDRA and on the Program Compound Case Retrieval The most recent Compound Case Retrieval Strategy (CRS) at the time of database lock will be used to determine the MedDRA search criteria to identify events of special interests.

#### 2.8.2 Deaths

The primary reason for death will be summarized by system organ class and preferred term. All deaths will be listed.

## 2.8.3 Laboratory data

The summary of laboratory evaluations will be presented for three groups of laboratory tests: Hematology, Chemistry and Urinalysis.

The number and percentage of patients with newly occurring or worsening laboratory abnormalities meeting the clinically notable criteria at any post-baseline visit will be summarized by laboratory parameter. For a patient to meet the criterion of a newly occurring clinically notable value, the patient needs to have a baseline value that is not clinically notable for that parameter. For a patient to meet the criterion of a worsening clinically notable value, the patient needs to have a baseline value that is clinically notable and also have a worse post-baseline value. For patients with missing baseline value, any post-baseline notable value will be considered as newly occurring.

Incidence of newly occurring liver enzymes abnormalities and renal events will be summarized using the number and percentage of patients by treatment group. Notable laboratory values will be listed.

Laboratory assessements performed at the follow-up visits in the scope of the USM will not be included in the summaries but will be listed. That means, assessments reported 21 days after end of study date will not be included in the summary tables.

## **Liver function tests (LFT)**

To evaluate potential drug-induced liver injury, the number and percentage of patients with newly occurring or worsening abnormalities in liver function tests at any time post-baseline will be summarized by treatment. The same approach as for notable laboratory values will be used to define newly occurring or worsening abnormalities in liver function tests.

When a criterion contains multiple laboratory parameters, the criterion will only be considered to have been met when all conditions occur at the same time (i.e., within the same sample). A case where all criteria are met at a post-baseline time point will be considered as newly occurring if the criteria are not met at baseline and will be considered as worsening if the criteria are met at baseline and at least one component is worsening from baseline irrespective of whether the other(s) are better.

Listings of patients with clinically notable LFT values will be provided.

The same analysis will be repeated for the Treatment withdrawal epoch.

## 2.8.4 Other safety data

#### 2.8.4.1 ECG

The (uncorrected) QT interval will be corrected according to Fridericia's formulae. The incidence rates of newly occurring or worsening clinically notable ECG abnormalities will be summarized. The same approach as for notable laboratory values will be used to define a newly occurring notable QTc value and a worsening notable QTc value. Notable ECG values will be listed.

Notable criteria are:

- QTcF > 500 msec or
- increase from baseline > 60 msec

If the single ECG shows a QTcF > 500 ms (males or females), 2 additional ECG replicates should be recorded to confirm the safety findings and copies forwarded to the central ECG laboratory for assessment. The results from those triplicate ECGs will be averaged and analysed as one value for summary and notable tables.

# 2.8.4.2 Vital signs

The number and percentage of subjects with clinically notable vital signs will be presented. Notable vital sign values will be listed.

#### Notable criteria are:

| Variable | Criterion value | | Change relative to baseline |
|---|---|---|---|
| Heart rate/pulse | 120 bpm<br>50 bpm | and an and a | increase of ≥ 15 bpm<br>decrease of ≥ 15 bpm |
| Systolic blood pressure | 180 mm Hg<br>90 mm Hg | and an and a | increase of ≥ 20 mm Hg<br>decrease of ≥ 20 mm Hg |
| Diastolic blood pressure | 105 mm Hg<br>50 mm Hg | and an and a | increase of ≥ 15 mm Hg<br>decrease of ≥ 15 mm Hg |
| Weight | Baseline weight (kg) | and an and a | increase of ≥ 7% decrease of ≥ 7% |

bpm= beats per minute

Data of subjects with newly occurring notable vital signs abnormalities will be listed in an additional listing.

#### 2.8.4.3 Physical examination

Physical examination including examination of skin will be source documentation only.



# 2.9 Pharmacokinetic endpoints

Scatter plots of EMA401 plasma concentrations will be displayed in linear and semilogarithmic view in a CSR addendum or in a separate report.

# 2.10 PD and PK/PD analyses

Evaluation of effect of EMA401 exposure on efficacy variables (e.g. change from baseline of pain score), via the development of a continuous descriptive Pharmacokinetics/ Pharmacodynamics (PK/PD) was planned in the protocol. All population PK/PD analyses and simulations were to be carried out using a non-linear mixed-effects modelling approach. Due to early study termination the planned model based exposure-response analysis will not be performed and replaced with a graphical assessment of the exposure-response relationship.

This will be reported in a separate report.

# 2.11 Patient-reported outcomes

Please refer to efficacy analysis for details on all Patient Reported Outcomes (PRO).

#### 2.12 Biomarkers

Not applicable.



# 2.14 Interim analysis - Safety

The DMC will review cumulative safety data, including patient narratives for deaths, serious adverse events (SAEs), discontinuations due to adverse events and cases of interest (allergic dermatitis, and clinically significant abnormal hepatic and hematology values).

The details of the analysis required for DMC will be specified in a separate DMC analysis plan and not repeated here in detail.

# 3 Sample size calculation

The calculation of power for the testing procedure mentioned in Figure 2-1 is based on the following assumptions:

- The treatment difference of 100 mg b.i.d. vs. placebo was assumed as 0.7, 0.8 and 0.9 points, for the primary efficacy variable (weekly mean of the 24-hour average pain score). A treatment difference of 0.7 points was observed for the 100 mg b.i.d. dose vs. placebo for weekly mean of the 24-hour average pain score (NRS) in the Study EMA401-003 during a 4-week treatment period. The standard deviation is 2.6 points (based on data from pregabalin historical trials see FDA Approval Package Medical Review, 2004) is assumed for the primary efficacy variable. In Study EMA401-003 in PHN patients, a standard deviation of approximately 2.0 points was observed. A slightly higher value of 2.6 has been chosen to account for a possible higher variability due to a higher number of centers and due to multiple imputations (as opposed to single imputation) in the analysis. It is also assumed that the same standard deviation holds for the PDN population.
- Treatment differences of 5 points for Pregabalin and 10 points for Duloxetine on NPSI total score were observed via an indirect comparison using the results from Tesfaye (2013) which is an active control study (Pregabalin vs Duloxetine) and Kalliomäki (2013) which is a placebo controlled study (AZD2423 vs placebo). The standard deviation was derived as 16 points using the results from Kalliomäki (2013). A correlation of approximately 0.2 was observed between the baseline scores of NRS and NPSI total score in Freeman et al (2014). The power of the study was calculated assuming correlation coefficient values of 0 and 0.2. Since the power values obtained for correlation values of 0.2 and 0 are similar, in a conservative scenario the results reported herein are for correlation value of 0.

Since the NPSI has not been studied in the EMA401-003 study, to mitigate the risk of uncertainty on the value of treatment difference and standard deviation, the effect size (treatment difference/ standard deviation) of NPSI total score has been considered for the calculation of power. The power of the study was calculated for different effect sizes ranging in 0.1, 0.5 for NPSI total score corresponding to 100 mg.

Under the assumptions of a 0.8 point treatment difference between 100 mg b.i.d. and placebo, a standard deviation as 2.6 for the primary efficacy variable and an effect size of 0.4 for 100

mg b.i.d. for the key secondary variable, N=200 patients per treatment arm will provide approximately 85% power to show that 100 mg b.i.d. is statistically significant over placebo for the primary efficacy variable, using the testing procedure mentioned in Figure 2-1. The power of showing the statistical significance of 100 mg b.i.d. dose in terms of the key secondary variable will be 84% under the same scenario. If we assume the treatment difference of 0.7 for the NRS as observed in the 4-week PoC study and the effect size for NPSI as 0.35, then the power for the primary objective will be 77% and that for the key secondary objective will be 72%. If the treatment difference between 100 mg b.i.d. and placebo is 0.9 for the NRS, and effect size is 0.45 for 100 mg b.i.d. for the NPSI, the power increases to 94% for the primary objective. The corresponding power for the key secondary objective increases to 93%.

# 4 Change to protocol specified analyses

An additional population, the mFAS population, has been defined.

The following analyses were specified in the protocol but will not be performed due the early termination of study:

- first and third supplementary analysis to the primary analysis
- tipping point analysis
- supplementary responder analyses
- ANCOVA analyses for BPI-SF, worst NRS pain score, ISI,
- proportional odds model for PGIC
- analyses regarding maintenance effect of EMA401 over placebo
- time to "sustained" pain reduction
- Apart from analyses of clinical abnormalities summaries of laboratory data, vital signs and ECG intervals have been removed
- Shift tables of laboratory data
- No safety figures will be presented
- Bazett correction for QTc



The following analyses have been added:

- sensitivity analyses on modified full analysis population
- analyses of TEAEs with onset before study termination date

The analyses of patient disposition for the treatment and treatment withdrawal epoch will be based on the FAS population only

Analyses of duration of exposure to study treatment will be based on the SAF population only.

Due to the early study termination only a few patients has been included in the region 'America'. To avoid convergence problems the covariate region has been removed from the ANCOVA model and from the logistic regression.

# 5 Appendix

# 5.1 Imputation rules

#### 5.1.1 Study drug

Missing/partial start date or end date of study treatment will not be imputed.

## 5.1.2 Diagnosis of PDN

Rules for imputing date of first diagnosis of PDN will be provided in Programming Dataset Specification (PDS) document in details.

#### 5.1.3 AE date imputation

Rules for imputing AE end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

## 5.1.4 Concomitant medication date imputation

Rules for imputing the CM end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

#### 5.1.5 Prohibited medication for PDN

Exclusion period of values in case of changed PDN medication or intake of prohibited medication will be derived as follows:

- Programming Dataset Specification (PDS) will describe how to identify dose changes of concomitant PDN medications and prohibited medications
- deterimine exclusion period: CM end date + x days where x=3 for changes in dose and x=7 for intake of prohibited medications with potential confounding effect
- if no medication end date available, then all values from medication start date onwards should be excluded

# 5.2 AEs coding/grading

The MedDRA version which will be available at the time of database lock, will be used for the coding purpose of the adverse events.

# 5.3 Laboratory parameters derivations

Liver events defined by laboratory parameter abnormalities (additional non-lab criteria as provided in the protocol are ignored):

- ALT or AST  $> 5 \times ULN$
- $ALP > 2 \times ULN$
- $TBL > 2 \times ULN$
- ALT or AST  $> 3 \times ULN$  and INR > 1.5
- ALT or AST >  $3 \times$  ULN and TBL >  $2 \times$  ULN AND ALP  $\leq 2 \times$  ULN (Potential Hy's Law cases)
- ALT or AST  $> 3 \times ULN$

Renal events defined by laboratory parameter abnormalities (additional non-lab criteria as provided in the protocol are ignored):

- Serum creatinine increase 25 49% compared to baseline
- Serum creatinine increase  $\geq 50\%$  compared to baseline
- New dipstick proteinuria ≥1+
- New dipstick glycosuria  $\ge 1+$  not due to diabetes
- New dipstick hematuria ≥1+ not due to trauma
- Albumin- or Protein-creatinine ratio increase >2-fold
- Albumin-creatinine ratio (ACR)  $\geq$ 30 mg/g or  $\geq$ 3 mg/mmol
- Protein-creatinine ratio (PCR) ≥150 mg/g or >15 mg/mmol

Laboratory results will be reported in SI units.

### 5.4 Derivation of index values and scores

For details on handling of missing items and derivation of scores refer to the document "Handling of missing items and derivation of total scores". The most recent version of this document stored at

available before the database lock will be used as reference.

# 5.4.1 11-point Numeric Rating Scale (NRS)

The Numeric Rating Scale (NRS) is an 11-point scale for patient self-reporting of pain. The averaged score will be computed for every week, regardless of visits.

#### 24-hour Average Pain Score

The 24-hour average pain score will be assessed using the 11-point numeric rating scale (NRS) scale ranging from zero to ten.

#### 24-hour Worst Pain Score

The 24-hour worst pain score will also be assessed using the 11-point NRS scale ranging from zero to ten.

## 5.4.2 Verbal Rating Scale (VRS) pain intensity

The Verbal Rating Scale (VRS) is a questionnaire administered by the clinician to capture the patient's level of pain. The response will be recorded as 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The score is recorded at baseline only.

## 5.4.3 Brief Pain Inventory- Short Form (BPI-SF)

Patients will be asked to complete the 7-item pain interference scale which assesses the degree to which pain interferes with walking and other physical activity, work, mood, relations with others and sleep using a zero to ten numeric rating scale, with zero being "does not interfere" and ten being "completely interferes". The score is recorded at Visits 101, 104, 106, 199, TD visit.

The BPI interference total score will derived as the sum of the 7 responses for the questions 9A-9G. The total score ranges from 0 to 70.

## 5.4.4 Patient Global Impression of Change (PGIC)

The Patient Global Impression of Change (PGIC) is a patient-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse"). The score is recorded at Visit 199 and TD visit only.

## 5.4.5 Neuropathic Pain Symptom Inventory (NPSI)

The Neuropathic Pain Symptom Inventory (NPSI) is a 12 item patient reported outcome measure that contains 10 descriptors representing 5 dimensions of pain (burning pain, deep/pressing pain, paroxysmal pain, evoked pain and paraesthesia/dysesthesia) and 2 temporal items designed to assess pain duration and the number of pain paroxysms. The score is recorded at Visits 101, 104, 106, 199, 201 and TD visit.

The sum of the responses to the 10 questions (all except qn. 4 and qn. 7) will be regarded as the total score and will be used for the analysis.

The dimensional score of each of the five dimensions are calculated as follows:

- Burning = Q1
- Pressing = (Q2 + Q3)/2
- Paroxysmal = (Q5 + Q6)/2
- Evoked = (O8 + O9 + O10)/3
- Paraesthesia / dysesthesia = (Q11 + Q12)/2

# 5.4.6 Insomnia Severity Index (ISI)

Patients will be asked to complete the ISI using five-point Likert-style scale as a measure of perceived sleep difficulties. Scores can range from zero to 28, with a cut-off score of eight suggesting the presence of sub-threshold insomnia. The questionnaire assesses the severity of insomnia, satisfaction with current sleep pattern, sleep interference, "noticeability" of sleeping problem to others and concern about sleeping problems. The score is recorded at Visits 101, 199 and TD visit.

The sum of seven responses represents the total score. Each of the 7 items is scored using a range from 0 to 4, thus the total score values can range from zero to 28.



For business use only

Novartis

Page 33

# 5.4.12 Douleur Neuropathique 4 (DN4)

The Douleur Neuropathique 4 (DN4) is a clinician administered questionnaire that can be useful in diagnosing neurophatic pain (Bouhassira et al 2005). DN4 consists of 10 items. Seven items are related to pain quality and are based on an interview with the patient, and 3 items are based on the clinical examination. This score is recorded at Screening only. Each of the 10 items has a dichotomous answer Yes (=1) or No (=0). The global score is calculated as the sum of the 10 items.

#### 5.5 Statistical models

SAS codes for all statistical methodology described in this section will be included as programming note in TFL Shells.

## 5.5.1 Primary analysis

#### 5.5.1.1 ANCOVA

The primary analysis (and all other analyses of continuous variables) will be done using analysis of covariance. The model is:

mean pain score = intercept + treatment + sex + age + PDNmed (yes/no) + baseline (mean pain intensity) + error.

The SAS procedure MIXED will be used for computing p-values and 95% confidence intervals for LS means.

#### 5.5.1.2 Missing data imputation

For the purpose of missing data imputation, the following two scenarios will be considered:

- Jump to reference (J2R)
- Missing At Random (MAR)

The imputation will be based on all available data (i.e. from all scheduled time points) using all covariates as specified in the ANCOVA model. For J2R only placebo data will be used, for MAR data from the same treatment arm will be used for building the imputation model.

#### 5.5.2 Secondary analysis

#### 5.5.2.1 Logistic regression

The proportion of responders will be analyzed using a repeated measures logistic regression. The model is similar to the ANCOVA model:

Response = intercept + treatment + sex + age + PDNmed (yes/no) + baseline (mean pain intensity) + error.

The SAS procedure GENMOD will be used.

Odds ratios will be presented along with 95% confidence intervals and p-values for the treatment contrasts.

## 5.6 Rule of exclusion criteria of analysis sets

Rule of exclusion criteria from analysis sets due to protocol deviations will be included prior to database lock.

## 6 References

Bouhassira D, Attal N, Alchaar H, et al (2005) Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain; 114(1-2):29-36.

Bretz F, Maurer W, Brannath W, et al (2009) A graphical approach to sequentially rejective multiple test procedures. Stat Med; 28(4):586-604.

Carpenter JR, Roger JH, Kenward MG (2013) Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat; 23(6):1352-71.

CEMA401A Handling of missing items in the derivation of total scores for efficacy measures (last version available before DB lock is used)

CEMA401A Estimand charter (last version available before DB lock is used)

CEMA401A Visit Windows for Baseline and Post-baseline visits and Treatment Discontinuation (TD) visit mapping (last version available before DB lock is used)

Freeman R, Baron R, Bouhassira D, et al (2014) Sensory profiles of patients with neuropathic pain based on the neuropathic pain symptoms and signs. Pain; 155(2):367–76.

Kalliomäki J, Attal N, Jonzon B, et al (2013) A randomized, double-blind, placebo-controlled trial of a chemokine receptor 2 (CCR2) antagonist in posttraumatic neuralgia. Pain; 154(5):761-67.

Permutt T (2015) Sensitivity analysis for missing data in regulatory submissions. Stat Med; 35:2876-9

Pinheiro J, Bornkamp B, Glimm E, et al (2014) Model-based dose finding under model uncertainty using general parametric models. Statist Med; 33:1646–61.

Markus et. al. (1976), On closed testing procedures with special reference to ordered analysis of variance, Biometrika (1976), 63, 3 pp 655-60